CLINICAL TRIAL: NCT00846794
Title: Can AcuGraph Differentiate Between Participants With and Without Digestive Symptoms
Brief Title: AcuGraph and Digestive Symptoms
Status: Completed | Type: Observational
Sponsor: Logan College of Chiropractic (Other)
Responsible Party: Principal Investigator, Brian Snyder, DC, Research Associate, Logan College of Chiropractic
Other Study IDs: SR1219080169; 400
Record Dates: First submitted 2009-02-12; First posted 2009-02-19 (Estimated); Last update posted 2016-09-15 (Estimated); Status verified 2016-09

CONDITIONS: Digestive Disorders; Irritable Bowel Syndrome; Constipation; Diarrhea
MeSH Terms: conditions — Digestive System Diseases; Irritable Bowel Syndrome; Constipation; Diarrhea

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1 Asymptomatic: students with conditions being studied
- 2 Symptomatic: students without conditions being studied

SUMMARY:
This research is designed to study the reliability of the results of an AcuGraph in college students and faculty members with reported digestive symptoms

DETAILED DESCRIPTION:
The specific aim of the study is to test the reliability of the AcuGraph in subjects with irritable bowel syndrome (IBS). The hypothesis is that the AcuGraph will be a reliable method to identify disorders in subjects.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be required to answer a questionnaire evaluating for a percentage of digestive disorders "disability" based on the subject's answers. If a participant's answers do not qualify as a disability, they will be assigned to the asymptomatic group and will still be examined with an AcuGraph to provide normative data.

Exclusion Criteria:

* heart condition
* kidney disorder
* thyroid disorders
* diabetes
* chronic disease or illness
* neurological diseases
* skin or bleeding disorders
* pregnant
* currently taking drugs or nutritional supplements
* pacemaker and/or

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Logan students currently enrolled
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2009-02; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
AcuGraph: computerized device to analyze & document the energetic status of the acupuncture meridians | At examination

SECONDARY OUTCOMES:
IBS Questionnaire | At examination

CONTACTS AND LOCATIONS:
Locations (1):
- Logan University, College of Chiropractic, Chesterfield, Missouri, United States